CLINICAL TRIAL: NCT03629145
Title: The Effect of Live Music Therapy Interventions With Pediatric Patients Who Are Mechanically Ventilated and Sedated
Brief Title: Music Therapy With Intubated and Sedated Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Hannah Ivey, Music Therapist, Board-Certified, Children's Healthcare of Atlanta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUSIC02
Record Dates: First submitted 2017-11-21; First posted 2018-08-14 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live Music Therapy (Experimental): Twenty minutes of live, preferred music played on guitar and voice
  Interventions: Behavioral: Live Music Therapy
- Recorded Music (Placebo Comparator): Twenty minutes of recorded music, also on guitar and voice, previously recorded by investigator
  Interventions: Behavioral: Recorded Music Therapy

INTERVENTIONS:
Behavioral: Live Music Therapy — Investigator will begin play live guitar and voice music.
  Arms: Live Music Therapy
Behavioral: Recorded Music Therapy — Investigator will play recorded music.
  Arms: Recorded Music

SUMMARY:
The study is a randomized controlled trial of pediatric patients ages birth to two years of age who are mechanically ventilated and sedated as a result of a respiratory virus. The experimental group will receive twenty minutes of live, preferred music with a board-certified music therapist and the control group will receive twenty minutes of recorded music, also preferred, both interventions conducted at bedside. Caregivers will take a pre and post survey.

DETAILED DESCRIPTION:
Data for heart rate, respiratory rate, and blood pressure will be taken for both control and experimental conditions prior to intervention, immediately following intervention, thirty minutes post, and sixty minutes post intervention. Caregivers will take the Parental Belief Scale for Hospitalized Children prior to intervention and 60 minutes poster intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory syntactical virus, pneumonia, rhino, corona, bronchiolitis, or flu
* mechanically ventilated
* sedated
* Patients with underlying diagnosis accepted unless listed below
* Patients must have a primary caregiver present

Exclusion Criteria:

* Patients who are oscillating
* have a previous diagnosis of severe or profoundly deaf
* have a suspicion of child abuse
* in custody of the state.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate | up to sixty minutes post intervention.
  Describe the effect of a live music therapy intervention on HR in patients ages 0 to 2 years who are mechanically ventilated and sedated in one PICU.
Respiratory Rate | up to sixty minutes post intervention.
  Describe the effect of a live music therapy intervention on RR in patients ages 0 to 2 years who are mechanically ventilated and sedated in one PICU.
Blood Pressure | up to sixty minutes post intervention.
  Describe the effect of a live music therapy intervention on BP in patients ages 0 to 2 years who are mechanically ventilated and sedated in one PICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin D. The psychophysiological effects of music therapy in intensive care units. Paediatr Nurs. 2010 Apr;22(3):14-20. doi: 10.7748/paed2010.04.22.3.14.c7637. PMID 20426353
- [Result] Han L, Li JP, Sit JW, Chung L, Jiao ZY, Ma WG. Effects of music intervention on physiological stress response and anxiety level of mechanically ventilated patients in China: a randomised controlled trial. J Clin Nurs. 2010 Apr;19(7-8):978-87. doi: 10.1111/j.1365-2702.2009.02845.x. PMID 20492042
- [Result] Hetland B, Lindquist R, Chlan LL. The influence of music during mechanical ventilation and weaning from mechanical ventilation: A review. Heart Lung. 2015 Sep-Oct;44(5):416-25. doi: 10.1016/j.hrtlng.2015.06.010. Epub 2015 Jul 27. PMID 26227333

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03629145/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03629145/ICF_001.pdf